CLINICAL TRIAL: NCT02620319
Title: Biodegradable Stents in the Management of Stenoses of the Large Airways
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol turned out to be not quite suitable for most patients. Apart from Thomayer's hospital, 2 other centers could not cooperate. The introduction of stents continued at the Thomayer Hospital. Publication of results is planned in 2024.
Sponsor: Ludek Stehlik (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); University Hospital Olomouc (Other); University Hospital, Motol (Other)
Responsible Party: Sponsor-Investigator, Ludek Stehlik, MUDr., Thomayer University Hospital
Organization: Thomayer University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT 14146-3/2013; NT14146 (Other Grant/Funding Number: Internal Grant Agency of the Czech Ministry of Health)
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Tracheal Stenosis
Keywords: bronchoscopy; polydioxanone; absorbable implants; stents
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- biodegradable stent (Experimental): endoscopic implantation of biodegradable airway stent, the SX-ELLA Stent DV Tracheal (DV Stent)
  Interventions: Device: SX-ELLA Stent DV Tracheal (DV Stent)

INTERVENTIONS:
Device: SX-ELLA Stent DV Tracheal (DV Stent) — The trachea is intubated with a rigid bronchoscope while participants are placed under total intravenous anesthesia and jet ventilation. The delivery apparatus containing the stent is introduced through a rigid tube to the desired depth under visual control. Then the stent is deployed and its position is determined and, if necessary, stent is repositioned using rigid forceps. In-stent balloon dilation is carried out. If needed, thoracic surgeon can secure the stent in place via external (percutaneous) fixation: one suture is passed through the stent, the tracheal wall, soft tissues, and skin; the suture is then knotted on the skin of the neck. The suture is removed two to three weeks after implantation.
  Other Names: DV Stent

SUMMARY:
The objective of this project is to determine whether biodegradable polydioxanone stents are efficient in the treatment of adult patients with tracheobronchial stenoses.

DETAILED DESCRIPTION:
Background:

The ideal airway stent has yet to be developed. Biodegradable (BD) stents are made of knitted polymer fibers that degrade when placed in the body; extraction of the device is, therefore, unnecessary. Several in vitro and in vivo studies of tracheal BD stents composed of various materials have been conducted.

Polydioxanone is a biodegradable polymer in the polyester family, which has attracted a lot of interest due to its exquisite biocompatibility and is currently available on the market in the form of absorbable suture material. It is degraded by hydrolysis (of its ester bonds), which is accelerated under low potential of Hydrogen (pH) conditions, into harmless degradation products. Polydioxanone tracheal stents appear to be well tolerated by the tracheal mucosa, retain their mechanical strength for as long as 6 weeks, and, in animal models, completely degrade after approximately 15 weeks. They have been successfully used in humans as mechanical support for tracheal transplants, during treatment of obstructive airway complications after lung transplantation, and in children with airway stenosis.

Hypotheses:

Biodegradable stents can be used in adult patients as a temporary mechanical support of narrowed airways, they allow healing of the airways or secure the airways until another (anticancer, anti-inflammatory) therapy manages the cause of the narrowing. Biodegradable stents are expected to have advantages over classical stents, namely good biocompatibility, fair adaptation to the anatomy of the airways, they do not limit the transportation of secretions substantially.

Objectives:

The primary objective of this study is to show that BD stents can be safely used and are effective in the treatment of adult patients with tracheal narrowings.

The secondary objectives are: to observe and analyze mucosa - BD stent interaction, to assess degradation of stents and its consequences.

Design:

Prospective interventional study conducted in three hospitals in the Czech Republic.

Methods:

The investigators intend to enroll adult participants suffering from significant large airway stenoses in which the stenting is generally considered to be effective. Every participant is reviewed by at least two interventional pulmonologists and a thoracic surgeon to determine the best therapeutic option. Bronchoscopy and computed tomography of the trachea is considered essential to confirm the diagnoses. All participants sign an informed consent form prior to undergoing the procedure.

During the stent implantation, the trachea is intubated with a rigid bronchoscope, participants are placed under total intravenous anesthesia and jet ventilation. The investigators intend to use self-expandable, biodegradable, polydioxanone tracheal stents, the SX-ELLA Stent DV Tracheal (DV Stent), manufactured by ELLA-CS, s.r.o., Hradec Kralove, Czech Republic. Stent is standardly equipped with radiopaque markers at distal and proximal end. It is delivered in sterile packed, separately from original delivery system into which the stent immediately before implantation is placed. As mentioned, stent is made of synthetic polymer - braided polydioxanone fiber widely used for absorbable surgical suture. The suture has successfully been used in the surgery, orthopedics and dental surgery for more than 25 years. It is known that the material is subjected to the bulk hydrolytic degradation in the body. No toxic substances arise within the degradation process. The ultimate degradation substance is 2-hydroxyacetic acid that is finally metabolized to water and carbon dioxide. The data about local reaction produced by polydioxanone implants, incl. buried sutures are contradictory. Majority of them report very low tissue reaction.

The first bronchoscopy follow up is carried out during the first post-implantation week, additional follow-ups (including clinical evaluation, bronchoscopy, basic spirometry, and chest X-ray if needed) are performed on a monthly or as-needed basis. If the restenosis threatens, the participant can be given another polydioxanone stent, as well as, he or she can be treated using mechanical removal of obstacles, balloon dilation, laser therapy and electrocautery.

Results are analyzed continuously, final evaluation is intended to be performed after reaching a sufficient number of participants. This includes statistical analysis of overall results in participants after complete stent degradation, assessment of major clinical signs and functional parameters, and especially, evaluations of endoscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* significant large airway stenoses
* benign tracheobronchial stenosis of any origin in participants who can not go for surgery, or who refuse surgical treatment
* benign tracheobronchial stenoses of any origin when the surgery is planed after some delay, benign tracheobronchial stenoses when the effect of anti- inflammatory or anti-infective treatment is expected
* malignant tracheobronchial stenoses due to extrinsic compression when exhausted curative modalities
* malignant stenoses from extrinsic compression in participants undergoing the actinotherapy or receiving systemic anticancer therapy

Exclusion Criteria:

* stenoses of any origin which can be treated primarily surgically
* stenoses caused by intraluminal growth of tumor, tracheoesophageal or bronchoesophageal fistulas
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
airway patency during the presence of the stent in the airways | residence time of the stent in the airways, i.e. as long as no stent material is found, up to 180 days after implantation, since then the stent is not considered to provide any mechanical support
  Scheduled bronchoscopies, trachea is, for the purposes of the study, classified according to Freitag's recommended adapted classification system (Freitag L. et al. A proposed classification system of central airway stenosis, Eur Respir J 2007; 30:7-12).

SECONDARY OUTCOMES:
number of complications: infection, bleeding, migration, obstructive granulation tissue formation, sudden restenosis (of any origin, unexpected in relation to the degree of the stent degradation) | residence time of the stent in the airways (i.e. as long as no stent material is found, up to 180 days after implantation, since then the stent is not considered to provide any mechanical support) and 6 months thereafter
evaluation of forced expiratory volume in 1 second (FEV1) | residence time of the stent in the airways (i.e. as long as no stent material is found, up to 180 days after implantation, since then the stent is not considered to provide any mechanical support) and 6 months thereafter
  FEV1 (in liters and % predicted values) measurements within follow-ups.
evaluation of forced vital capacity (FVC) | residence time of the stent in the airways (i.e. as long as no stent material is found, up to 180 days after implantation, since then the stent is not considered to provide any mechanical support) and 6 months thereafter
  FVC (in liters and % predicted values) measurements within follow-ups.
airway patency after complete degradation of the stent or loss of majority support functions | six months, beginning after identifying the complete degradation of the stent or 180 days after implantation
  Scheduled bronchoscopies, trachea is, for the purposes of the study, classified according to Freitag's recommended adapted classification system (Freitag L. et al. A proposed classification system of central airway stenosis, Eur Respir J 2007; 30:7-12).

CONTACTS AND LOCATIONS:
Overall Officials: Ludek Stehlik, MUDr., Principal Investigator — Department of Respiratory Medicine, Thomayer Hospital, Videnska 800, 140 59 Praha 4; Miloslav Marel, Prof. MUDr., Study Director — Department of Pneumology, 2nd Faculty of Medicine, Charles University in Prague and Motol University Hospital; Vitezslav Kolek, Prof. MUDr., Study Director — Department of Respiratory Diseases and Tuberculosis, University Hospital Olomouc; Martina Vasakova, Prof. MUDr., Study Director — Department of Respiratory Medicine, Thomayer Hospital, Videnska 800, 140 59 Praha 4
Locations (3):
- Czechia (3):
  - Department of Respiratory Diseases and Tuberculosis, University Hospital Olomouc, Olomouc
  - Department of Respiratory Medicine, Thomayer Hospital, Prague
  - Department of Pneumology, 2nd Faculty of Medicine, Charles University in Prague and Motol University Hospital, Prague

REFERENCES:
- [Background] Novotny L, Crha M, Rauser P, Hep A, Misik J, Necas A, Vondrys D. Novel biodegradable polydioxanone stents in a rabbit airway model. J Thorac Cardiovasc Surg. 2012 Feb;143(2):437-44. doi: 10.1016/j.jtcvs.2011.08.002. Epub 2011 Aug 31. PMID 21885070
- [Background] Lischke R, Pozniak J, Vondrys D, Elliott MJ. Novel biodegradable stents in the treatment of bronchial stenosis after lung transplantation. Eur J Cardiothorac Surg. 2011 Sep;40(3):619-24. doi: 10.1016/j.ejcts.2010.12.047. Epub 2011 Feb 21. PMID 21334911
- [Background] Vondrys D, Elliott MJ, McLaren CA, Noctor C, Roebuck DJ. First experience with biodegradable airway stents in children. Ann Thorac Surg. 2011 Nov;92(5):1870-4. doi: 10.1016/j.athoracsur.2011.07.042. Epub 2011 Oct 31. PMID 22051281
- [Background] Chin CS, Litle V, Yun J, Weiser T, Swanson SJ. Airway stents. Ann Thorac Surg. 2008 Feb;85(2):S792-6. doi: 10.1016/j.athoracsur.2007.11.051. PMID 18222219
- [Background] Korpela A, Aarnio P, Sariola H, Tormala P, Harjula A. Bioabsorbable self-reinforced poly-L-lactide, metallic, and silicone stents in the management of experimental tracheal stenosis. Chest. 1999 Feb;115(2):490-5. doi: 10.1378/chest.115.2.490. PMID 10027451
- [Background] Korpela A, Aarnio P, Sariola H, Tormala P, Harjula A. Comparison of tissue reactions in the tracheal mucosa surrounding a bioabsorbable and silicone airway stents. Ann Thorac Surg. 1998 Nov;66(5):1772-6. doi: 10.1016/s0003-4975(98)00763-2. PMID 9875787
- [Background] Saito Y, Minami K, Kobayashi M, Nakao Y, Omiya H, Imamura H, Sakaida N, Okamura A. New tubular bioabsorbable knitted airway stent: biocompatibility and mechanical strength. J Thorac Cardiovasc Surg. 2002 Jan;123(1):161-7. doi: 10.1067/mtc.2002.118503. PMID 11782770
- [Background] Freitag L, Ernst A, Unger M, Kovitz K, Marquette CH. A proposed classification system of central airway stenosis. Eur Respir J. 2007 Jul;30(1):7-12. doi: 10.1183/09031936.00132804. Epub 2007 Mar 28. PMID 17392320
- [Result] Hytych V, Horazdovsky P, Stehlik L, Pracharova S, Pohnan R, Lefnerova S, Vasakova M. Our own method of fixation of biodegradable tracheal stent. Bratisl Lek Listy. 2015;116(5):340-2. doi: 10.4149/bll_2015_064. PMID 25924646
- [Result] Stehlik L, Hytych V, Letackova J, Kubena P, Vasakova M. Biodegradable polydioxanone stents in the treatment of adult patients with tracheal narrowing. BMC Pulm Med. 2015 Dec 21;15:164. doi: 10.1186/s12890-015-0160-6. PMID 26690793
- [Result] Stehlik L, Guha D, Anandakumar S, Taskova A, Vasakova MK. Biodegradable tracheal stents: our ten-year experience with adult patients. BMC Pulm Med. 2024 May 15;24(1):238. doi: 10.1186/s12890-024-03057-y. PMID 38750487